CLINICAL TRIAL: NCT07140484
Title: A Single-arm, Open-label Phase IV Study to Evaluate the Effectiveness of Sotatercept in Improving Pulmonary Vascular Recruitment in Patients With Pulmonary Arterial Hypertension (PAH)
Brief Title: Sotatercept in Pulmonary Arterial Hypertension
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Merck Canada Inc. (Industry); Alberta Health services (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00148970
Record Dates: First submitted 2025-08-08; First posted 2025-08-24 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Pulmonary Artery Hypertension
Keywords: diffusing capacity; membrane diffusing capacity; pulmonary capillary blood volume
MeSH Terms: conditions — Familial Primary Pulmonary Hypertension | interventions — ACE-011

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Sotatercept Group (Experimental): Sotatercept 0.7mg/kg
  Interventions: Drug: Sotatercept

INTERVENTIONS:
Drug: Sotatercept — 0.7mg/kg
  Other Names: Winrevair

SUMMARY:
The goal of this clinical trial is to determine whether sotatercept is effective in improving diffusing capacity in patients with pulmonary arterial hypertension.

Participants will be asked to:

* Take Sotatercept every 21 days (±3 days)
* Each participant will be enrolled in the study for 29 Weeks
* Visit the clinic 18 times
* Have a physical exam
* Perform assessments of lung function and exercise tests
* Have an ultrasound of their heart
* Have blood draws done at regular intervals

The main objectives of the study are:

Primary objective: To assess whether sotatercept will improve recruitment of diffusing membrane capacity (DM) with exercise.

Secondary objective: To identify components of the diffusing capacity that respond to treatment with sotatercept in pulmonary arterial hypertension.

DETAILED DESCRIPTION:
Potential participants must provide their written informed consent before any study-specific procedures.

All screening procedures will be completed over two weeks during three separate visits. For participants from the Calgary site (site 2), all Visit 1 procedures except for PFT and CPET may be performed on a separate day in Calgary. Visits 2 and 3 will be performed in Edmonton (site 1). According to patient preference, visits 2 and 3 can be performed on the same day, with a minimum 3-hour break between visits. For participants from Calgary (site 2), the first drug administration will occur in Calgary within seven days of completion of Visit 3 procedures.

Screening will include reviewing the participant's medical, surgical, and family history, collecting demographics, race, and ethnicity, and requesting medical records for relevant external procedures.

Screening procedures include:

Visit 1:

* Informed consent
* Inclusion/exclusion criteria
* Medical history review
* Physical examination
* 12-lead ECG
* Vital signs
* Weight
* WHO FC assessment
* 6MWT
* Pregnancy test
* Hematology (complete blood count)
* Urinalysis
* Hemoglobin
* Serum chemistry
* NT-proBNP
* PFT
* CPET
* QoL assessments
* AE/SAE Review
* Concomitant medication review

Visit 2:

* Hemoglobin
* Rest/exercise DLCO, VC, DM
* Rest/exercise CW-NIRS
* AE/SAE Review
* Concomitant medication review

Visit 3:

* Pregnancy test
* Rest/exercise Echocardiography
* AE/SAE Review
* Concomitant Medication review
* Study drug administration

Measurements/assessments taken during the Screening Period will be recorded as the baseline values for the study assessment of endpoints.

Treatment Period (Visit 4-14) All study procedures should be performed prior to the study drug administration. For participants at the Calgary site, Visits 4,8-14 occur at their home site. For participants from the Calgary site (site 2), Visit 5-7 will be performed in Edmonton (site 1). Visits 5-7 are to be performed before the administration of the 3rd dose of the study drug. According to the patient's preference, visits 6 and 7 may be combined.

Visit 4 (Week 3)

* Focused cardiopulmonary physical examination
* Vital signs
* Weight
* WHO FC assessment
* 6MWT
* Pregnancy test
* Hematology
* Urinalysis
* Clinical worsening assessment
* AE/SAE Review
* Concomitant medication review

Visit 5 (Week 5-6):

* PFT
* CPET
* QoL assessments
* AE/SAE Review
* Concomitant medication review

Visit 6 (Week 5-6):

* Hemoglobin
* Rest/exercise DLCO, VC, DM
* Rest/exercise CW-NIRS
* AE/SAE Review
* Concomitant medication review

Visit 7 (Week 5-6):

* Pregnancy test
* Rest/exercise Echocardiography
* AE/SAE Review
* Concomitant Medication review

Visit 8 (Week 6):

* Focused cardiopulmonary physical examination
* 6MWT
* Vital signs
* Weight
* WHO FC assessment
* Pregnancy test
* Hematology
* Urinalysis
* Clinical worsening assessment
* AE/SAE Review
* Concomitant medication review

Visit 9 (Week 9):

* Focused cardiopulmonary physical examination
* 6MWT
* 12-lead ECG
* Vital signs
* Weight
* WHO FC assessment
* Pregnancy test
* Hematology
* Serum chemistry
* NT-proBNP
* Clinical worsening assessment
* AE/SAE Review
* Concomitant medication review

Visit 10-14 (Week 12 - 24):

* Focused cardiopulmonary physical examination
* 6MWT
* Vital signs
* Weight
* WHO FC assessment
* Pregnancy test
* Hematology
* Urinalysis
* Clinical worsening assessment
* AE/SAE Review
* Concomitant medication review

End-of-Study Period (Visits 13-14) End-of-Study period visits will start 1 week after the last dose of the study medication and will be completed over 2 weeks. Visits 15-17 will be performed in Edmonton (site 1). Visit 16 and 17 can be performed on the same day according to patient preference.

Visit 15:

* Weight
* Hemoglobin
* PFT
* CPET
* QoL Assessment
* AE/SAE Review
* Concomitant medication review

Visit 16:

* Hemoglobin
* Rest/exercise DLCO, VC, DM
* Rest/exercise CW-NIRS
* AE/SAE Review
* Concomitant medication review

Visit 17:

* Rest/exercise echocardiography
* AE/SAE Review
* Concomitant medication review

Follow-up period (Visit 18) A follow-up visit will occur 3 weeks after the last dose of the study medication. For Edmonton participants (site 1), Visit 18 may happen on the same day after Visit 17 is completed.

Visit 18:

* 6MWT
* 12-lead ECG
* Vital signs
* WHO FC assessment
* Pregnancy test
* Hematology
* Urinalysis
* NT-proBNP sample collection
* Clinical worsening assessment
* AE/SAE Review
* Concomitant medication review

Following the last dose of study drug administration, participants have the option to continue with open label sotatercept supplied directly from the manufacturer until either the participant discontinues sotatercept or reimbursement through public or private insurance is in place. The treating physician will be responsible for ongoing monitoring and administration of sotatercept beyond the last dose.

ELIGIBILITY:
Eligible participants must meet all of the following inclusion criteria to be enrolled in the study:

1. Age ≥ 18 years.
2. Documented diagnostic right heart catheterization (RHC) at any time prior to screening confirming the diagnosis of PAH Group 1 in any of the following subtypes:

   * Idiopathic PAH
   * Heritable PAH
   * Drug/toxin-induced PAH
   * PAH associated with CTD
   * PAH associated with simple, congenital systemic-to-pulmonary shunts at least 1 year following repair.
3. Symptomatic PAH classified as WHO FC II or III.
4. On stable doses of ≥2 background PAH therapies for at least 60 days prior to screening; for infusion prostacyclins, dose adjustment within 10% of the optimal dose is allowed per medical practice. Patients on 1 background PAH therapy are eligible if there is documented intolerance or contraindication to use of the other 2 classes (e.g. liver enzyme elevation while taking an ERA).
5. Females of childbearing potential must:

   * Have a negative urine or serum pregnancy tests as verified by the investigator prior to starting study therapy.
   * If sexually active, have used, and agree to use highly effective contraception without interruption during the study (including dose interruptions), and for 16 weeks (112 days) after discontinuation of study treatment.
   * Refrain from breastfeeding a child or donating blood, eggs, or ovum for the duration of the study and for at least 16 weeks (112 days) after the last dose of study treatment.
6. Male participants must:

   * Agree to use a condom, defined as a male latex condom or nonlatex condom NOT made out of natural (animal) membrane (e.g., polyurethane), during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions and for at least 16 weeks (112 days) following investigational product discontinuation, even if he has undergone a successful vasectomy.
   * Refrain from donating blood or sperm for the duration of the study and for 16 weeks (112 days) after the last dose of study treatment
7. Ability to adhere to study visit schedule and understand and comply with all protocol requirements.
8. Ability to understand and provide written informed consent.

Exclusion Criteria

1. 1. Diagnosis of pulmonary hypertension WHO Groups 2, 3, 4, or 5
2. Musculoskeletal limitation that precludes participation in cycle ergometry
3. Resting oxygen saturation < 88%. (Note: patients on oxygen can be included in the study if they can maintain a resting saturation of ≥ 88 % after 3 minutes off oxygen).
4. Diagnosis of the following PAH Group 1 subtypes: human immunodeficiency virus (HIV)-associated PAH and PAH associated with portal hypertension, schistosomiasis-associated PAH and pulmonary veno-occlusive disease.
5. Hemoglobin (Hgb) at screening above the gender-specific upper limit of normal (ULN), per local laboratory test.
6. Baseline platelet count < 50,000/mm3 (< 50.0 × 109/L) in the enrollment period.
7. Uncontrolled systemic hypertension as evidenced by sitting systolic blood pressure > 160 mmHg or sitting diastolic blood pressure > 100 mmHg during a screening visit after a period of rest.
8. Baseline systolic blood pressure < 90 mmHg at screening.
9. Pregnant or breastfeeding women.
10. Any of the following clinical laboratory values at the screening visit:

    * Estimated glomerular filtration rate (eGFR) < 30 mL/min/m2 (as defined by the Modification of Diet in Renal Disease [MDRD] equation)
    * Serum alanine aminotransferase, aspartate aminotransferase, or total bilirubin levels > 3 × ULN (bilirubin criterion waived if there is a documented history of Gilbert's syndrome).
11. Currently enrolled in or have completed any other investigational product study within 30 days for small-molecule drugs or within 5 half-lives for biologics prior to the date of signed informed consent.
12. History of full pneumonectomy.
13. Pulmonary function test (PFT) values of forced vital capacity (FVC) < 60% predicted and/or FEV1/FVC < lower limit of normal at the screening visit or within 6 months prior to the screening visit.
14. Smoking history of ≥ 20 pack-years or any tobacco smoking or vaping within the previous 3 months.
15. Body mass index ≥ 40 kg/m2.
16. Planned initiation of an exercise program for cardiopulmonary rehabilitation during the study (participants who are stable in the maintenance phase of a program and who will continue for the duration of the study are eligible).
17. Known history of portal hypertension or chronic liver disease, including hepatitis B and/or hepatitis C (with evidence of recent infection and/or active virus replication), defined as mild to severe hepatic impairment (Child-Pugh Class A-C).
18. History of restrictive, constrictive, or congestive cardiomyopathy.
19. History of atrial septostomy within 180 days prior to the screening visit.
20. Electrocardiogram (ECG) with Fridericia's corrected QT interval (QTcF) > 500 ms during the Screening Period
21. Personal or family history of long QT syndrome (LQTS) or sudden cardiac death.
22. Left ventricular ejection fraction < 45% on historical echocardiogram within 6 months prior to the screening visit.
23. Any symptomatic coronary disease events (prior myocardial infarction, percutaneous coronary intervention, coronary artery bypass graft surgery, or cardiac anginal chest pain) within 6 months prior to the screening visit. Note: Anginal pain can be ignored as an exclusion criterion if coronary angiography shows no obstructions.
24. Cerebrovascular accident within 3 months prior to the Screening Visit.
25. Significant mitral or aortic valve dysfunction (greater than moderate mitral regurgitation or aortic regurgitation, or greater than mild mitral stenosis or aortic stenosis).
26. Received intravenous inotropes (e.g., dobutamine, dopamine, norepinephrine, vasopressin) within 30 days prior to the screening visit.
27. Known hypersensitivity to sotatercept or to any ingredient in the formulation or component of the container.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-10-06 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Lung diffusing capacity | 6 weeks post starting treatment
  Lung diffusing capacity (DLCO) will be measured using six-second, advanced DLCO techniques
Lung diffusing capacity | 23 weeks post starting treatment
  Lung diffusing capacity (DLCO) will be measured using six-second, advanced DLCO techniques
Diffusing membrane capacity (Dm) | 6 weeks post starting treatment
  Diffusing membrane capacity will be measured using six-second, advanced DLCO
Diffusing membrane capacity (Dm) | 23 weeks post starting treatment
  Diffusing membrane capacity will be measured using six-second, advanced DLCO
Pulmonary capillary blood volume (Vc) | 6 weeks post starting treatment
  Pulmonary capillary blood volume (Vc) will be measured using six-second, advanced DLCO techniques
Pulmonary capillary blood volume (Vc) | 23 weeks post starting treatment
  Pulmonary capillary blood volume (Vc) will be measured using six-second, advanced DLCO techniques

SECONDARY OUTCOMES:
Cardiac structure and function | 6 weeks post starting treatment
  Cardiac structure will be measured using standard cardiac ultrasound
Cardiac structure and function | 23 weeks post starting treatment
  Cardiac structure will be measured using standard cardiac ultrasound
Cardiac function | 6 weeks post starting treatment
  Cardiac function will be measured using standard cardiac ultrasound
Cardiac function | 23 weeks post starting treatment
  Cardiac function will be measured using standard cardiac ultrasound
Peripheral muscle microcirculation | 6 weeks post starting treatment
  Peripheral muscle microcirculation will be measured using continuous-wave near-infrared spectroscopy
Peripheral muscle microcirculation | 23 weeks post starting treatment
  Peripheral muscle microcirculation will be measured using continuous-wave near-infrared spectroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Jason Weatherald, MD, Principal Investigator — University of Alberta; Michael Stickland, PhD, Principal Investigator — University of Alberta
Locations (1):
- Clinical Physiology Laboratory, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No